CLINICAL TRIAL: NCT06134102
Title: Clinical and Laboratory Characteristics of Polycythemia Vera
Acronym: PV-ARC
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 483/2018/Oss/AOUBo
Record Dates: First submitted 2023-10-05; First posted 2023-11-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2023-02

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is observational, longitudinal, retrospective and prospective, on patients with PV. Patients with PV diagnosed from 2000 to 2023 according to WHO2017 criteria will be considered. The main purpose of the study is to determine the impact of clinical and laboratory characteristics of Polycythemia Vera on patients' prognosis, understood as long-term survival

DETAILED DESCRIPTION:
The structured collection of data necessary for the evaluation of the objectives will take place through the creation of a specific electronic archive with an expected duration of 7 years, possibly extendable. The electronic archive may be used to review case histories and to obtain or confirm new scientific evidence on Polycythemia Vera. Patients will be followed and treated within the care pathway provided by normal clinical practice.

The following elements will be considered in each patient: age, recent and remote pathological history, characteristics of PV onset, histological, cytogenetic and molecular investigations of diagnostic definition, medical therapies performed, type of response to the therapies performed, complications of these therapies and pathology. All useful data will be collected exclusively through consultation of outpatient medical records.

The planned enrollment period is 60 months (January 2019-December 2023). The observation period of enrolled patients is at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PV according to WHO 2017 criteria,
* Obtaining informed consent for data collection and processing

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The incidence of PV is approximately 11 x 1,000,000 patient-years. For the purpose of the registry, clinical/laboratory data collection will be expanded to 22 Hematology Centers experienced in the study of chronic myeloproliferative neoplasms. Overall, about 150 new diagnoses per year are expected from all Centers. Considering that about 20 percent of patients will not be able to be included for various reasons (lack of diagnosis according to WHO2017 criteria, patient's failure to refer to Hematology Centers, refusal to participate in the study), the registry is expected to include clinical data from about 2000 cases diagnosed from 2000 to the year 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Long-term survival | 6 years
  To determine the impact of clinical and laboratory characteristics of Polycythemia Vera (PV) on patients' prognosis, in terms of lon term survival

SECONDARY OUTCOMES:
Thrombosis | 6 years
  To assess the incidence of thrombotic events on PV patients
Haemorrhages | 6 years
  To assess the incidence of haemorrhagic events on PV patients
Therapies | 6 years
  To assess the use of high-cost therapies
Therapies Toxicity | 6 years
  To assess the toxicity of therapies
Therapies Efficacy | 6 years
  To assess the effects of therapies
Development of second neoplasms | 6 years
  To assess the incidence of second malignancies
Evolution to acute leukemias | 6 years
  To assess the incidence of acute leukaemias

CONTACTS AND LOCATIONS:
Locations (22):
- Italy (22):
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Apulia
  - Grande Ospedale Metropolitano "Bianchi Melacrino Morelli", Reggio Calabria, Calabria
  - IRCCS Policlinico Sant'Orsola, Bologna, Emilia-Romagna
  - Università degli studi di Ferrara - Nuovo Polo Ospedaliero di Cona - A.O.U. Arcispedale S. Anna, Ferrara, Emilia-Romagna
  - Policlinico di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Parma, Parma, Emilia-Romagna
  - AUSL di Piacenza - Palazzine Medicine Specialistiche, Piacenza, Emilia-Romagna
  - Dipartimento Oncoematologico - AUSL della Romagna, Ravenna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia, Emilia-Romagna
  - Ospedale Infermi Rimini, Rimini, Emilia-Romagna
  - A.O.U. Integrata di Udine, Udine, Friuli Venezia Giulia
  - A.O.U. Policlinico Umberto I - Università degli Studi di Roma "La Sapienza", Rome, Lazio
  - IRCCS Azienda Ospedaliera Universitaria "San Martino" - IST, Genoa, Liguria
  - IRCCS per l'oncologia -Ospedale Policlinico "San Martino", Genoa, Liguria
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - A.O.U. Città della Salute e della Scienza - Presidio Molinette, Turin, Piedmont
  - Ospedale "A. Businco" - Dipartimento Scienze Mediche e Sanità Pubblica Università degli Studi di Cagliari, Cagliari, Sardinia
  - A.O.U. "Policlinico-V. Emanuele"- P.O. Ferrarotto, Catania, Sicily
  - A.O. Ospedali Riuniti Marche Nord - Presidio Ospedaliero San Salvatore, Pesaro, The Marches
  - AOU di Padova, Padua, Veneto
  - A.O.U. Integrata Verona - Borgo Roma, Verona, Veneto